CLINICAL TRIAL: NCT02119962
Title: A Working Memory Training in Burnout Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: HSK (Unknown)
Responsible Party: Principal Investigator, Ingmar Franken, Professor, Erasmus Medical Center
Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2014-04-08; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Burnout
Keywords: burnout; working memory; working memory training; cognitive behavioral therapy; executive control
MeSH Terms: conditions — Burnout, Psychological

ARMS (2):
- Working memory training (Experimental)
  Interventions: Behavioral: Working memory training
- Placebo training (Placebo Comparator)
  Interventions: Behavioral: Placebo training

INTERVENTIONS:
Behavioral: Working memory training
  Arms: Working memory training
Behavioral: Placebo training
  Arms: Placebo training

SUMMARY:
Burnout patients show deficient working memory functioning. Several studies showed a training can increase working memory capacity. In the current study we explored whether training working memory can reduce burnout and burnout related symptoms and increase working memory capacity.

ELIGIBILITY:
Inclusion Criteria:

* undifferentiated somatoform disorder with a work related cause

Exclusion Criteria:

* age which exceeded the range of 18 to 67 years
* a severe major depressive episode
* substance dependence or abuse

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-06; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change in Utrechtse Burnout Scale (UBOS) score on pre and post training and two months after training | Baseline, post (4 weeks after baseline), after last session of cognitive behavioral therapy and follow-up (2 months after post-test)
  The Dutch translation of the Maslach Burnout Inventory - General Survey (Schaufeli, Leiter, Maslach, & Jackson, 1996), the Utrechtse Burnout Scale-A, measures the severity of burnout symptoms.

SECONDARY OUTCOMES:
Change in Cognitive Failure Questionnaire (CFQ) score on pre and post training and two months after training | Baseline, post (4 weeks after baseline), after last session of cognitive behavioral therapy and follow-up (2 months after post-test)
  The Cognitive Failure Questionnarie measures the frequency of participants' experienced cognitive failures regarding memory, action, perception and attention.

OTHER OUTCOMES:
Change in Symptom Checklist-90-Revised (SCL-90) score on pre and post training and two months after training | Baseline, post (4 weeks after baseline), after last session of cognitive behavioral therapy and follow-up (2 months after post-test)
  The Dutch version of the Symptom Checklist-90-Revised (Derogatis, 1977) is a 90-item self-report questionnaire which measures psychosocial distress of the last week - including the day of testing - on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely).
Change in Digit Span score on pre and post training and two months after training | Baseline, post (4 weeks after baseline), after last session of cognitive behavioral therapy and follow-up (2 months after post-test)
  The Digit Span consists of two parts with 14 trials each: the forward Digit Span measures short term memory, whereas the backward version measures WM.
Change in Reading Span partial-credit unit score on pre and post training and two months after training | Baseline, post (4 weeks after baseline), after last session of cognitive behavioral therapy and follow-up (2 months after post-test)
  The Reading Span assesses the processing and storage functions of WM (Shipstead et al., 2012).

CONTACTS AND LOCATIONS:
Locations (1):
- HSK, Arnhem, Gelderland, Netherlands